CLINICAL TRIAL: NCT02850042
Title: Comparing Constraint-Induced Therapy and Occupation-Based Intervention for Optimal Stroke Recovery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lumy Sawaki (Other)
Responsible Party: Sponsor-Investigator, Lumy Sawaki, Associate Professor,department of Physical Medicine and Rehabilitation, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-0509
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Stroke; Cerebrovascular Accident
Keywords: motor recovery; human; occupation-based practice; motor training; transcranial magnetic stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Occupation-based practice (Experimental): Occupation-based intervention (OBP) is a form of activity-based therapy consisting of client-directed occupations that match client-identified goals. OBP group will participate in activities such as wood working, scrap booking, higher level dressing (don/doffing a bra, zipping coat), hair care, opening doors, using bathroom stalls, typing, cooking, tying shoes, washing dishes, carrying dirty dish carts, clearing dirty dishes and raking. Repetition of the tasks are not the focus in the OBP group. Each session lasted 55-minute and it was delivered twice a week for 4 weeks (8 sessions).
  Interventions: Behavioral: Occupation-based practice (OBP)
- Modified-constraint induced therapy (Active Comparator): Modified-constraint induced therapy (m-CIT) group will target functional goals (eg, activities of daily living) or goal subcomponents (eg, pinching, grasp/release, or functional reach patterns). Tasks were repeated at rate of approximately 10 to 50 repetitions each session according to the demands of the task. No physical constraint of the less-affected UE will be applied, but training compelled highly repetitive use of the more-affected upper extremity. Subjects will attempt tasks with progressive difficulty. Each session lasted 55-minute and it was delivered twice a week for 4 weeks (8 sessions).
  Interventions: Behavioral: Modified-constraint induced therapy (m-CIT)

INTERVENTIONS:
Behavioral: Occupation-based practice (OBP)
  Arms: Occupation-based practice
Behavioral: Modified-constraint induced therapy (m-CIT)
  Arms: Modified-constraint induced therapy

SUMMARY:
This pilot study was designed to compare the effects of modified constraint-Induced therapy and occupation-based intervention to increase functional motor recovery in stroke

DETAILED DESCRIPTION:
The purpose of this study is to investigate change in motor performance and the extent of neuroplastic change associated with both occupation-based intervention and modified constraint-Induced therapy (m-CIT) in the recovery of upper extremity motor function following a stroke. Transcranial Magnetic Imaging (TMS) will be used to compare the difference in the brain reorganization of each client before and after the intervention to identify which technique is more effective in changing brain function. Central Hypothesis: Stroke subjects with motor deficit receiving occupation-based interventions will demonstrate improved motor function greater to that of the subjects receiving m-CIT interventions. Sixteen participants with chronic stroke will be recruited for the study over the age 21. Participants will be randomly assigned to one of the two therapy groups and will receive 55 minutes of therapy 2 times per week for 4 weeks for a total of 8 sessions.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age and older
* at least 12 months from stroke
* mild-to-severe upper extremity motor deficit
* single ischemic or hemorrhagic stroke

Exclusion Criteria:

* history of head injury with loss of consciousness
* seizures
* severe alcohol or drug abuse
* psychiatric illness interfering with participation in the study including uncontrolled depression
* cognitive deficits severe enough to preclude informed consent
* ferromagnetic material near the brain
* individuals that could be pregnant
* cardiac or neural pacemakers
* if currently receiving occupational therapy services

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assessment (FMA | Score change after 8 days of intervention compared to baseline

SECONDARY OUTCOMES:
Stroke Impact Scale (SIS) | Score change after 8 days of intervention compared to baseline
Canadian Occupational Performance Measure (COPM) | Score change after 8 days of intervention compared to baseline
Goal Attainment Scale (GAS). | Score change after 8 days of intervention compared to baseline
Transcranial Magnetic Stimulation (map volume) | Score change after 8 days of intervention compared to baseline

IPD SHARING:
Plan to Share IPD: Undecided